CLINICAL TRIAL: NCT02797054
Title: Culturally Tailored Educational Intervention to Improve Decision Quality Around Humanpapillomavirus (HPV) Vaccination
Brief Title: Educational Intervention to Improve HPV Vaccination Decision Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 14-0402-1
Record Dates: First submitted 2016-05-31; First posted 2016-06-13 (Estimated); Results first posted 2018-08-24 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-08

CONDITIONS: HPV Vaccination Decision Quality
Keywords: HPV vaccination; Vaccination decision-making; Tailored health messaging; Barriers to vaccination; Attitudes
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tailored Intervention (Experimental): Intervention: tailored educational materials. In this arm, participants will complete a baseline survey on an iPad, view a series of educational webpages on the iPad, and complete a brief post intervention survey.
  Interventions: Behavioral: Tailored educational materials
- Untailored Intervention (Other): Intervention: untailored educational materials. In this arm, patients will view educational information on the iPad that is not responsive to their baseline questionnaire answers.
  Interventions: Behavioral: Untailored educational materials
- Usual Care (Other): Intervention: usual care as experienced during appointment with primary care provider. Participants in the usual care arm will not view any educational materials or complete the baseline survey.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Tailored educational materials — The tailored intervention will use participants' baseline survey responses to generate tailored educational messages about the HPV vaccine. These educational messages will reflect the top concerns indicated by the participant about the HPV vaccine. Additional tailoring will occur in the form of images matched to self-reported race and age, and using participants' first name in the information presented.
  Arms: Tailored Intervention
Behavioral: Untailored educational materials — The untailored intervention will present educational information on the iPad that is not responsive to participants' baseline questionnaire answers and instead is derived directly from the HPV "Vaccine Information Sheet" that has been created by the Centers for Disease Control and Prevention.
  Arms: Untailored Intervention
Behavioral: Usual care — Those in the usual care arm will be provided with a paper version of the Post Intervention Survey. This will be provided to participants after their clinic visit is completed.
  Arms: Usual Care

SUMMARY:
The purpose of this study is to evaluate an innovative approach to improving HPV vaccination among the Hispanic population. The objectives/aims of this HPV educational intervention project are:

1. To measure the quality of the HPV vaccine decision among participants in different arms of the intervention
2. To determine patterns of intervention utilization among participants in different arms of the intervention, and

The implementation of this educational intervention in clinic waiting rooms is intended to assist primary care providers in communicating HPV vaccine awareness and education to parents and patients in a culturally tailored format.

DETAILED DESCRIPTION:
While HPV infection is nearly ubiquitous among the sexually active population, the morbidity and mortality from HPV-related diseases disproportionately affects minorities and the poor. Hispanic women are at particularly high risk as they have the highest rates of invasive cervical cancer when compared to all other racial or ethnic groups in the U.S. Initiating the 3-dose HPV vaccination series is more common among Hispanic adolescents than whites, but series completion has been lowest among Hispanic populations.

To understand barriers to HPV vaccination and to provide insight into ways in which an existing educational intervention should be modified for a Hispanic population, the investigators conducted focus groups among Hispanic parents and Latina young adults. All groups reported vaccine cost, access to insurance, and a general lack of awareness and/or understanding of either HPV or the vaccine as barriers. All groups also wanted substantially more "general" information about both HPV and the vaccine in order to make informed vaccination decisions. The educational intervention was generally well received but there were universal suggestions from all the groups to provide additional basic information about HPV infection, to add information about the vaccine for boys/young men, and to modify the color scheme and logo to make it more eye-catching and pleasing.

This current phase of the project will be comprised of real world testing of an iPad-based educational intervention about HPV, "Combatting HPV Infection and Cancer" (CHICOS) that has been revised and developed per focus group feedback to target the Hispanic population.

By providing information that patients and parents have clearly indicated they want in a way that is culturally sensitive and meaningful and also individually personalized, the investigators hope to improve the HPV vaccination decision-making process.

ELIGIBILITY:
Inclusion Criteria:

1. Parents of an adolescent between the ages of 9-17
2. A young adult patient between the ages of 18-26
3. Adolescent/young adult who has not yet received all three doses of the HPV vaccine.
4. Parent/young adult who can read and converse in either English or Spanish

Exclusion Criteria:

1. Age <18,
2. Prisoners
3. Decisionally challenged subjects
4. Those who cannot read and converse in either English or Spanish
5. Those who have received all 3 doses of the HPV vaccine

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1205 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda F Dempsey, MD, PhD, MPH, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Post-test
Arm/Group | Tailored Intervention | Untailored Intervention | Usual Care
Started | 387 | 383 | 435
Completed | 380 | 372 | 87
Not Completed | 7 | 11 | 348
Period: Follow-up
Arm/Group | Tailored Intervention | Untailored Intervention | Usual Care
Started (All participants who volunteered at consent were contacted for follow-up.) | 387 | 383 | 435
Completed | 178 | 155 | 150
Not Completed | 209 | 228 | 285

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tailored Intervention | Untailored Intervention | Usual Care | Total
Number analyzed (Participants) | 387 | 383 | 435 | 1205
Age, Customized [Mean (Full Range); unit: Years]
  Age | 32.01 [18 to 59] | 31.18 [17 to 55] | 31.60 [17 to 60] | 31.60 [17 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 386 | 382 | 434 | 1202
  Male | 1 | 1 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 349 | 342 | 392 | 1083
  Not Hispanic or Latino | 36 | 41 | 40 | 117
  Unknown or Not Reported | 2 | 0 | 3 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 88 | 98 | 105 | 291
  Race: African American | 4 | 1 | 2 | 7
  Race: Asian | 2 | 1 | 0 | 3
  Race: American Indian | 6 | 6 | 6 | 18
  Race: Other | 285 | 277 | 319 | 881
  Race: Unknown | 2 | 0 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants - Who Agreed They Felt Sure About the Best Choice Regarding the HPV Vaccine at Post-intervention
Time Frame: 1 day
Measure: Number; unit: Percent of participants
Arm/Group | Tailored Intervention | Untailored Intervention | Usual Care
Number analyzed (Participants) | 380 | 372 | 87
Percent of participants | 94 | 95 | 89
Statistical Analysis 1: Comparison: Tailored Intervention vs Untailored Intervention vs Usual Care; Test type: Other; p = 0.069, Chi-squared

2. Primary Outcome: Percent of Participants Who Agreed They Knew Enough About the Risks and Benefits of the HPV Vaccine at Post-intervention
Time Frame: 1 day
Measure: Number; unit: Percent of participants
Arm/Group | Tailored Intervention | Untailored Intervention | Usual Care
Number analyzed (Participants) | 380 | 372 | 87
Percent of participants | 75 | 77 | 69
Statistical Analysis 1: Comparison: Tailored Intervention vs Untailored Intervention vs Usual Care; Test type: Other; p = 0.303, Chi-squared

3. Primary Outcome: Percent of Participants Who Agreed They Felt Clear About Which Risks and Benefits of the HPV Vaccine Mattered Most to Them at Post-intervention
Time Frame: 1 day
Measure: Number; unit: Percent of participants
Arm/Group | Tailored Intervention | Untailored Intervention | Usual Care
Number analyzed (Participants) | 380 | 372 | 87
Percent of participants | 85 | 87 | 71
Statistical Analysis 1: Comparison: Tailored Intervention vs Untailored Intervention vs Usual Care; Test type: Other; p = 0.001, Chi-squared

4. Primary Outcome: Percent of Participants Who Agreed They Felt They Had Enough Support to Make a Decision About Getting the HPV Vaccine at Post-intervention
Time Frame: 1 day
Measure: Number; unit: Percent of participants
Arm/Group | Tailored Intervention | Untailored Intervention | Usual Care
Number analyzed (Participants) | 380 | 372 | 87
Percent of participants | 86 | 87 | 86
Statistical Analysis 1: Comparison: Tailored Intervention vs Untailored Intervention vs Usual Care; Test type: Other; p = 0.895, Chi-squared

5. Primary Outcome: Percent of Participants Who Agreed They Felt Sure About the Best Choice Regarding the HPV Vaccine at Follow-up
Time Frame: 2 Months
Measure: Number; unit: percent of participants
Arm/Group | Tailored Intervention | Untailored Intervention | Usual Care
Number analyzed (Participants) | 149 | 155 | 176
percent of participants | 96 | 95 | 94
Statistical Analysis 1: Comparison: Tailored Intervention vs Untailored Intervention vs Usual Care; Test type: Other; p = 0.58, Chi-squared

6. Primary Outcome: Percent of Participants Who Agreed They Knew Enough About the Risks and Benefits of the HPV Vaccine at Follow-up
Time Frame: 2 Months
Measure: Number; unit: Percent of participants
Arm/Group | Tailored Intervention | Untailored Intervention | Usual Care
Number analyzed (Participants) | 149 | 153 | 177
Percent of participants | 76 | 73 | 60
Statistical Analysis 1: Comparison: Tailored Intervention vs Untailored Intervention vs Usual Care; Test type: Other; p = 0.0015, Chi-squared

7. Primary Outcome: Percent of Participants Who Agreed They Felt Clear About Which Risks and Benefits of the HPV Vaccine Mattered Most to Them at Follow-up
Time Frame: 2 Months
Measure: Number; unit: Percent of participants
Arm/Group | Tailored Intervention | Untailored Intervention | Usual Care
Number analyzed (Participants) | 148 | 154 | 178
Percent of participants | 78 | 78 | 65
Statistical Analysis 1: Comparison: Tailored Intervention vs Untailored Intervention vs Usual Care; Test type: Other; p = 0.0056, Chi-squared

8. Primary Outcome: Percent of Participants Who Agreed They Felt They Had Enough Support to Make a Decision About Getting the HPV Vaccine at Follow-up
Time Frame: 2 Months
Measure: Number; unit: Percent of participants
Arm/Group | Tailored Intervention | Untailored Intervention | Usual Care
Number analyzed (Participants) | 150 | 155 | 176
Percent of participants | 85 | 84 | 77
Statistical Analysis 1: Comparison: Tailored Intervention vs Untailored Intervention vs Usual Care; Test type: Other; p = 0.21, Chi-squared

ADVERSE EVENTS:
Arm/Group | Tailored Intervention | Untailored Intervention | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/387 | 0/383 | 0/435
Other Adverse Events (participants affected / at risk) | 0/387 | 0/383 | 0/435

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No